CLINICAL TRIAL: NCT04528316
Title: Impact of Physical Activity on Postural Stability and Coordination in Children With Posterior Fossa Tumor
Brief Title: Physical Activity on Postural Stability and Coordination in Children With Posterior Fossa Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHE-BT003
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Posterior Fossa Tumor; Medulloblastoma, Childhood
Keywords: physical activity; postural stability; coordination; posterior fossa tumor
MeSH Terms: conditions — Infratentorial Neoplasms; Medulloblastoma; Motor Activity

STUDY DESIGN:
Intervention Model Description: Experimental controlled randomization using Block Stratified Randomized Software program, after obtaining informed consent from illegible patient or his caregiver.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group/Pilates Core Stability Exercises program Group (Active Comparator): Twenty patients will receive Pilates core stability exercises program ONLY. Total Period: 12 Weeks
  Stages: Three stages:
  * Stage I: Warm-up: consists of four Pilates motions:
    1. Breathing:
    2. Rolling back:
    3. Coccyx-curl:
    4. Hundred breathing:
  * Stage II: Work-out: consists of twelve Pilates motions:
    1. Single leg stretch:
    2. Straight leg raise:
    3. Basic bridge:
    4. Bridging variation:
    5. Quadruped:
    6. Clap with seal motion
    7. Mermaid twist:
    8. Swimming:
    9. Double leg stretch:
    10. Shoulder bridge:
    11. Swan dive:
    12. Leg full front:
  * Stage III: Cool-down: consists of three Pilates motions:
    1. Rest position:
    2. Cat with arm/leg extension:
    3. Breathing:
  Interventions: Behavioral: Pilates Core Stability Exercises program
- Balance Group (Experimental): Twenty patients will receive the same selected Pilates core stability exercises program given to control group in addition to Balance Program
  Interventions: Behavioral: Pilates Core Stability Exercises program; Behavioral: Balance Program
- Coordination Group (Experimental): Twenty patients will receive the same selected Pilates core stability exercises program given to control group in addition to Coordination Exercises.
  Interventions: Behavioral: Pilates Core Stability Exercises program; Behavioral: Coordination

INTERVENTIONS:
Behavioral: Pilates Core Stability Exercises program — Twenty patients will receive Pilates core stability exercises program ONLY. Total Period: 12 Weeks
  Stages: Three stages:
  * Stage I: Warm-up: consists of four Pilates motions:
    1. Breathing:
    2. Rolling back:
    3. Coccyx-curl:
    4. Hundred breathing:
  * Stage II: Work-out: consists of twelve Pilates motions:
    1. Single leg stretch:
    2. Straight leg raise:
    3. Basic bridge:
    4. Bridging variation:
    5. Quadruped:
    6. Clap with seal motion
    7. Mermaid twist:
    8. Swimming:
    9. Double leg stretch:
    10. Shoulder bridge:
    11. Swan dive:
    12. Leg full front:
  * Stage III: Cool-down: consists of three Pilates motions:
    1. Rest position:
    2. Cat with arm/leg extension:
    3. Breathing:
Behavioral: Balance Program — Total Period: 12 Weeks. The designed HUMAC program will work on the modified clinical test of sensory integration of balance (mCTSIB) with eyes open and with eyes closed, the center of pressure (COP) and the limit of stability test (LOS).
  Other Names: HUMAC program
  Arms: Balance Group
Behavioral: Coordination — Total Period: 12 Weeks. Coordination will be assessed using BOT2, Bilateral coordination (Sub test No.4) composed of 7 items and Upper-Limb coordination (Sub test No.7) composed of 7 items too.
  The raw scores are recorded first then it is converted into point scores, then subtest total point score is obtained by adding point scores.
  Arms: Coordination Group

SUMMARY:
Medulloblastoma is a rapidly-growing tumor of the cerebellum, this area controls balance, posture and sophisticated motor functions like finer hand movements, speech, and swallowing. It has been reported that those children fall frequently so the purpose of this study is to investigate the effectiveness of balance and coordination training in these Children.

DETAILED DESCRIPTION:
The effects of physical exercise training interventions for childhood cancer participants are not yet convincing due to small numbers of participants and insufficient study methodology. More and high-quality evidence is needed in order to be able to draft exercise and physical activity guidelines for this population. Despite the positive results of exercise interventions in adult cancer patients, the evidence for benefits in childhood cancer patients is limited.

There are Two Main objectives:

1. To investigate the effectiveness of Pilates core stability exercises program. 2. To investigate the effectiveness of Humac balance and tilt system.

Secondary Objectives:

1. The effectiveness of coordination training in children with posterior fossa tumors.
2. The comparison between balance and coordination training and which of both trainings has more effect.

This study will take place in a pediatric oncology setting, Children's Cancer Hospital Egypt(CCHE), in outpatient setting. Patients will be evaluated for their balance and coordination at initial presentation, during treatment, and during follow-up after end of treatment at CCHE. Also patients will receive balance and coordination training, before each chemotherapy cycle-maximum one week- given the patient is in good state.

Sixty children with posterior fossa tumors of both sexes will participate in this study. They will be selected from CCHE. They will be randomly assigned into 3 groups of equal number.

ELIGIBILITY:
Inclusion Criteria:

1. Children with posterior fossa tumors during follow up.
2. Children between 5-12 years old.
3. Time elapsed since the start of treatment more than 4 months in order to be in maintenance phase.
4. They can understand verbal command.
5. Children with no visual, auditory or perceptual disorders.
6. Children are already treated surgically.

Exclusion Criteria:

* Children who have one or more of the following criteria will be excluded from the study:

  1. Children with a genetic disorder or mental retardation.
  2. Children with a chronic lung disease.
  3. Sever cardiomyopathy (ejection fraction <40%, ischemia and angina pectoris at rest).
  4. Children with a neuromuscular disease not related to tumor.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change Balance | at week 12
  For assessment of the three groups, HUMAC balance and tilt system will be used to assess both Static and dynamic balance.

SECONDARY OUTCOMES:
Change Coordination | at week 12
  The Bruininks-Oseretsky Test of Motor Proficiency - Second Edition
  - The minimum and maximum values: Coordination will be assessed using BOT2, Bilateral coordination (Sub test No.4) composed of 7 items and Upper-Limb coordination (Sub test No.7) composed of 7 items too.
  The raw scores are recorded first then it is converted into point scores, then subtest total point score is obtained by adding point scores.
  Bilateral Coordination: Total Point Score Subtest (min=Zero, max=24). Upper-Limb Coordination: Total Point Score Subtest (min=Zero, max=39).
  - Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Usama Mahmoud Ahmed, MSc, Principal Investigator — Cairo University
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, Egypt

REFERENCES:
- [Derived] Usama M, Abdelaziem F, Rashed WM, Maher E, El Beltagy M, Zekri W. Impact of physical activity on postural stability and coordination in children with posterior fossa tumor: randomized control phase III trial. J Cancer Res Clin Oncol. 2023 Aug;149(9):5637-5644. doi: 10.1007/s00432-022-04490-4. Epub 2022 Dec 16. PMID 36525069